CLINICAL TRIAL: NCT00300495
Title: Phase III Study of Preoperative Amiodarone for Prevention of Atrial Fibrillation After Lung Resection
Brief Title: Study of Amiodarone Given Before Lung Surgery to Prevent Atrial Fibrillation After Lung Resection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to accrual total number of participants during study period.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Malcolm DeCamp, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005P000376
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation; Lung Cancer
Keywords: Atrial fibrillation; Lung cancer; Pulmonary resection; Post-operative complications
MeSH Terms: conditions — Atrial Fibrillation; Lung Neoplasms | interventions — Amiodarone; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 - Amiodarone (Experimental): Perioperative amiodarone
  Interventions: Drug: Amiodarone
- 2 - Control (Active Comparator): Control arm, standard care with no perioperative amiodarone
  Interventions: Other: Control arm, standard care

INTERVENTIONS:
Drug: Amiodarone — Perioperative orally administered
  Other Names: Cordarone; Pacerone
  Arms: 1 - Amiodarone
Other: Control arm, standard care — Control
  Arms: 2 - Control

SUMMARY:
Atrial fibrillation is a very common complication of pulmonary resection. Patients who develop atrial fibrillation require additional treatment and are more likely to stay in the hospital for longer period of time increasing the costs associated with the operation. We propose a randomized controlled trial to see if oral amiodarone given for one week before surgery can prevent atrial fibrillation after pulmonary resection. We plan to evaluate the incidence of atrial fibrillation in patients who received preoperative amiodarone and compare them to the incidence of atrial fibrillation in patients who did not received preoperative amiodarone.

DETAILED DESCRIPTION:
Atrial fibrillation is a very common complication of pulmonary resection. Patients who develop atrial fibrillation require additional treatment and are more likely to stay in the hospital for longer period of time increasing the costs associated with the operation.

We propose a study to see if oral amiodarone given for one week before surgery can prevent atrial fibrillation after pulmonary resection. We plan to evaluate the incidence of atrial fibrillation in patients who received preoperative amiodarone and compare them to the incidence of atrial fibrillation in patients who did not received preoperative amiodarone.

ELIGIBILITY:
Inclusion Criteria:

* Resectable lung nodule or mass

Exclusion Criteria:

* Allergy to amiodarone
* Currently taking amiodarone
* Documented atrial fibrillation within past 12 months
* Known pulmonary fibrosis
* Known hepatic dysfunction
* Thyroid disease
* 2nd or 3rd degree heart block
* Severe SA node disease
* Bradycardia-induced syncope
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2009-10-13 (Actual); Study Completion 2009-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm M DeCamp, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient in the control group was excluded because, after patient was enrolled, patient had mediastinoscopy that showed more advanced disease. Thus, patient did not undergo lung resection. Therefore this patient was excluded from the study.
Groups:
- 1 - Amiodarone: Perioperative amiodarone
  Amiodarone: Perioperative orally administered
  Patients received 200 mg of amiodarone three times a day for one week prior to surgery and 200 mg twice a day for one week after the surgery
Period: Overall Study
Arm/Group | 1 - Amiodarone | 2 - Control
Started | 10 | 9
Completed | 6 | 8
Not Completed | 4 | 1
Not completed — Protocol Violation | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Amiodarone | 2 - Control | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Customized [Count of Participants; unit: Participants]
  Age > 18 | 10 | 9 | 19
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-operative Atrial Fibrillation
Description: Number of patients with post-operative atrial fibrillation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1 - Amiodarone | 2 - Control
Number analyzed (Participants) | 6 | 8
Participants | 1 | 1

2. Secondary Outcome: Length of Post-operative Hospital Stay
Description: Length of hospital stay after the operation
Time Frame: 1 week on average
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 1 - Amiodarone | 2 - Control
Number analyzed (Participants) | 6 | 8
Days | 5 (2) | 5 (4)

ADVERSE EVENTS:
Time Frame: 1 week prior to surgery and 30 days after surgery
Arm/Group | 1 - Amiodarone | 2 - Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No